CLINICAL TRIAL: NCT03937778
Title: Sensory Afferents for Deep Pressure Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190089; 19-AT-0089
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Results first posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Normal Physiology
Keywords: Somatosensory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tourniquet block to left upper arm (Experimental): Participants underwent ~10 minutes of baseline testing followed by a tourniquet placement to left upper arm and inflated to 80-100 mmHG above systolic blood pressure. Participants repeatedly rated a variety of sensory stimuli after tourniquet was placed. Participants rated intensity and pleasantness of slow brushing and deep pressure on both hands/forearms at baseline and after loss of A-beta sensation.
  Interventions: Behavioral: Deep pressure block

INTERVENTIONS:
Behavioral: Deep pressure block — Apply deep pressure block by using blood pressure cuff.

SUMMARY:
Background:

Much is known about how people perceive light touch, temperature, and pain. But less is known about how deep pressure is perceived. Deep pressure is an important part of many touch therapies, like massage therapy. Researchers want to learn more to help people with chronic pain and other disorders.

Objective:

To find out which sensory nerve fibers are involved in feeling the sensation of deep pressure.

Eligibility:

Healthy people ages 18 50 enrolled in study number 16-AT-0077

Design:

Participants will be screened under study number 16-AT-0077

Participants will have 1 visit that lasts about 2 hours.

Participants will have a brief medical interview. They will have a urine test.

Participants will have ischemic nerve block on 1 arm. A blood pressure cuff will be inflated until the arm is numb for up to an hour.

Participants will have tests to see how they perceive different sensations. They will rate gentle brushing on the hands and forearms. They will rate gentle pressure squeezing from a hand massager on the hands and forearms.

Participants will receive other sensations such as vibration, cool, warm, pinprick without piercing the skin, finger movement, and pressure. They will be asked to rate or respond to the sensations. They will be asked to rate any pain or discomfort from the nerve block on an ongoing basis.

DETAILED DESCRIPTION:
Objective:

The sensory basis of non-painful deep pressure sensation is not known. We recently found that innocuous pressure sensation is eliminated in rare sensory neuronopathy patients with a specific loss of A-beta fibers, strongly suggesting that A-beta fibers underlie the ability to sense deep pressure. In addition, we and others have shown that deep pressure touch (observed in hugs and massage) frequently conveys a sense of pleasantness. The current study aims to examine the role of A-beta fibers in the perception of deep pressure touch including both its intensity and the pleasant affect it often elicits. This study constitutes the second study of the K99 phase of a K99/R00 grant application awarded to Dr. Laura Case by National Center for Complementary and Integrative Health (NCCIH).

Study Population:

Up to 24 healthy participants will be enrolled in the study with a goal of 12 completers. Participants will be invited based on previous screening and participation in our studies.

Design: Participants will undergo an ischemic-compression block. Sensory stimuli will be administered at frequent intervals to capture the loss of sensation related to A fibers as the block progresses. Before and after A-beta-associated sensations have been lost, the perception of deep pressure will be tested. Participants will rate the intensity and pleasantness of the pressure. Ratings of pain and discomfort will be collected throughout the study session.

Outcome measures: Primary outcome; Rating of intensity of deep pressure on the blocked arm before versus after loss of A-beta sensation, compared to ratings on the unblocked arm.

Secondary outcomes: 1) Rating of pleasantness of deep pressure on the blocked arm after loss of A-beta sensation, compared to ratings on the unblocked arm; 2) Ratings of intensity and pleasantness of gentle brushing on the blocked arm after loss of A-beta sensation, compared to ratings on the unblocked arm.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be:

* Between 18 and 50 years old.
* Fluent in English.
* Able to provide written informed consent.
* Enrolled in 16-AT-0077, Clinical and Scientific Assessment of Pain and Painful Disorders

EXCLUSION CRITERIA:

* Unable to comply with study procedures.
* Have used recreational drugs in the past 30 days.
* Pregnancy or breastfeeding.
* Congenital upper limb deficiency or amputation.
* Peripheral neuropathy, dermatological condition such as scars or burns, or has had a tattoo in the testing region within the previous four weeks that might influence cutaneous sensibility.
* Current chronic pain condition or has had chronic pain in the past year (painful condition lasting more than six months), including ongoing treatment with medications for neuropathic pain (e.g. gabapentin, tricyclic antidepressants, pregabalin, tramadol).
* Major medical condition, such as kidney, liver, cardiovascular (including blood clots, hypertension, preexisting cardiac arrhythmia, lymphadenopathy), autonomic, pulmonary, or neurological problems (e.g., seizure disorder) or a chronic systemic disease (e.g., diabetes) or Raynaud s disease.
* Personal history or first-degree family history of blood clots or clotting and circulatory disorders
* History of a seizures or first-degree family member with a seizure disorder
* High (>140/90) or low (<90/60) blood pressure
* Current and untreated diagnosis of major depression, post-traumatic stress syndrome, bipolar disorder, psychosis, anxiety or panic disorder, alcohol or substance use disorders
* History of fainting with blood draws
* Any medical counter-indications to the nerve blocks.
* Participant s arm unable to fit in inflated arm blood pressure cuff
* Participant has taken any pain medication other than an over-the-counter NSAIDs or acetaminophen within the last month or for more than one month on a continual basis within last six months.
* Used topical pain-relieving creams in the testing area within 24 hours of testing or non-steroidal anti-inflammatory drugs (NSAIDS), (e.g. aspirin, ibuprofen, acetaminophen, or naproxen) within 3 days of testing
* Recent use of medications that increase risk of seizures (e.g. antidepressant Wellbutrin or antipsychotic Haldol)
* NIH employees who are subordinates, relatives, or co-workers of the investigators, or NCCIH DIR employees.

EXCLUSION CRITERIA FOR INDIVIDUAL STUDY SESSION:

* Shows signs of alcohol withdrawal syndrome, or has behavioral signs of intoxication: will be excluded immediately and not have the possibility to reschedule their session.
* Used topical pain-relieving creams in the testing area (e.g. methylsalicylate, capsaicin) within 24 hours of testing or used non-steroidal anti-inflammatory drugs (NSAIDS, e.g. aspirin, ibuprofen), acetaminophen, or naproxen within 3 days of testing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Chesler, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-AT-0089.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tourniquet Block to Left Upper Arm
Started | 7
Completed | 5
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Unable to obtain loss of A-beta sensation prior to loss of C-fiber sensation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tourniquet Block to Left Upper Arm
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 2
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Arms in the Change of Pressure Intensity From Baseline to After Loss of A-beta Sensation
Description: Difference between left (blocked) and right (control) arms in the change from baseline to after loss of A-beta sensation from nerve block. Measurement of perceived pressure intensity was assessed using a visual analog scale ranging from "no sensation" (0) to "highest possible intensity" (100).
Time Frame: From baseline to after loss of A-beta sensation, within one-hour session
Population: All participants who completed all phases of the testing session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tourniquet Block to Left Upper Arm
Number analyzed (Participants) | 5
Units on a scale | -25.0 (19.65960325)

2. Secondary Outcome: Difference Between Arms in the Change of Pressure Pleasantness From Baseline to After Loss of A-beta Sensation
Description: Difference between left (blocked) and right (control) arms in the change from baseline to after loss of A-beta sensation from nerve block. Measurement of perceived pressure pleasantness was assessed using a visual analog scale ranging from "no sensation" (0) to "highest possible intensity" (100).
Time Frame: From baseline to after loss of A-beta sensation, within one-hour session
Population: All participants who completed all phases of the testing session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tourniquet Block to Left Upper Arm
Number analyzed (Participants) | 5
Units on a scale | -11.4 (10.85357084)

3. Secondary Outcome: Difference Between Arms in the Change of Brushing Intensity From Baseline to After Loss of A-beta Sensation
Description: Difference between left (blocked) and right (control) arms in the change from baseline to after loss of A-beta sensation from nerve block. Measurement of perceived brushing intensity was assessed using a visual analog scale ranging from "no sensation" (0) to "highest possible intensity" (100).
Time Frame: From baseline to after loss of A-beta sensation, within one-hour session
Population: All participants who completed all phases of the testing session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tourniquet Block to Left Upper Arm
Number analyzed (Participants) | 5
Units on a scale | -18.6 (23.67065694)

4. Secondary Outcome: Difference Between Arms in the Change of Brushing Pleasantness From Baseline to After Loss of A-beta Sensation
Description: Difference between left (blocked) and right (control) arms in the change from baseline to after loss of A-beta sensation from nerve block. Measurement of perceived brushing pleasantness was assessed using a visual analog scale ranging from "no sensation" (0) to "highest possible intensity" (100).
Time Frame: From baseline to after loss of A-beta sensation, within one-hour session
Population: All participants who completed all phases of the testing session
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tourniquet Block to Left Upper Arm
Number analyzed (Participants) | 5
Units on a scale | -12.4 (16.07171428)

ADVERSE EVENTS:
Time Frame: One day within a one-hour session
Arm/Group | Tourniquet Block to Left Upper Arm
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03937778/Prot_SAP_000.pdf